CLINICAL TRIAL: NCT00358423
Title: Pilot Study of the Effect of Pegaptanib Sodium in Patients With Chronic, Post-Operative Cystoid Macular Edema
Brief Title: The Effect of Macugen in Patients With Chronic, Post-Operative Cystoid Macular Edema
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling eligible subjects
Sponsor: Johns Hopkins University (Other)
Collaborators: Eyetech Pharmaceuticals (Industry)
Responsible Party: Diana V. Do, MD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00001702
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Cystoid Macular Edema
Keywords: CME; Pegaptanib; Post-Surgical Ocular Inflammation
MeSH Terms: conditions — Macular Edema | interventions — pegaptanib

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Pegaptanib Sodium
- B (Placebo Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Pegaptanib Sodium — 0.3 mg/0.1 ml intravitreal injection, every 6 weeks, up to a total of 3 injections
  Other Names: Macugen
  Arms: A
Drug: Control — Sham injections, every 6 weeks, up to a total of 3 sham injections
  Arms: B

SUMMARY:
This research is being done to look at the effects of an experimental drug called pegaptanib (also called Macugen) for the treatment of swelling in the retina (the light sensitive tissue in the back of the eye) that can occur after cataract surgery. Swelling in the retina can lead to blurry vision.

The only treatment available for this condition is eye drops that decrease swelling in the back of the eye, but eye drops may not decrease the swelling in everyone. We want to see if pegaptanib can decrease swelling in the retina and improve vision in patients with swelling after cataract surgery.

DETAILED DESCRIPTION:
While only 1% to 2% of people following cataract surgery develop visual acuity loss from chronic post-surgical cystoid macular edema (CME), this represents approximately 20,000 individuals in the U.S. each year, and many more throughout the world. No current drug or surgical treatment is very effective in the management of chronic post-surgical CME. Topical non-steroidal anti-inflammatory medications, such as ketorolac drops 4 times a day (qid) for 3 months, have been shown to reduce the extent of fluorescein leakage on angiography in patients with this condition; however, compliance can be difficult, not all cases resolve following this treatment, the drop is not approved for this indication, and it is unknown if this treatment has an effect that lasts beyond 3 to 6 months. The fluorescein angiographic findings and the effects of ketorolac drops suggest that the condition is a result of increased permeability from inflammation and might resolve with a therapy that decreases abnormal vessel permeability. Recent studies have shown that vascular endothelial growth factor (VEGF) plays a major role in vessel permeability. Pegaptanib (Macugen) is an FDA-approved drug for wet AMD. Pegaptanib is a selective VEGF antagonist that blocks the effects of VEGF; therefore,pegaptanib may decrease vessel permeability and possibly decrease CME. Pegaptanib has been shown to have some activity in reducing retinal blood vessel leakage in diabetic patients with chronic macular edema (Macugen Diabetic Retinopathy Study Group. A phase II randomized double-masked trial of pegaptanib, an anti-vascular endothelial growth factor aptamer, for diabetic macular edema. Ophthalmology 2005;112:1747-57.), further supporting the hypothesis that it might be effective in other causes of chronic macular edema. We plan to conduct a pilot study of the effects of pegaptanib (up to 3 treatments of pegaptanib given as often as every 6 weeks for up to 12 weeks) in subjects with chronic post-surgical CME. If pegaptanib treatment is shown to be beneficial for this condition, additional studies could be performed to prove long-term effectiveness in patients with chronic CME or even for prophylaxis for patients known to be at high risk of developing CME following ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults (ages 18 years or older)
* Best corrected visual acuity < 20/40 but no worse than 20/800 in the study eye
* Best corrected visual acuity better than or equal to 20/200 in the fellow eye
* Post-surgical CME in the study eye as documented on OCT (central subfield >/= 250 microns)
* Women of child-bearing potential who are interested in participating in this study will use two effective forms of contraception prior to initiation of pegaptanib and then throughout the remainder of the study. For women of childbearing potential, results from a urine pregnancy test will be obtained prior to each injection with pegaptanib. Urine samples will be disposed of after the test is performed.
* Initiation of pegaptanib or sham injections may begin following at least 12 weeks of topical therapy for CME after cataract surgery or the other eye,if the best-corrected visual acuity has not improved by at least 5 letters and if the center point thickening on OCT has not improved by at least 20%. Patients who have been on topical ketorolac for greater than 12 weeks are still eligible for this study.

Exclusion Criteria:

* History of intravitreal steroid (triamcinolone) injection into the study eye or fellow eye within 4 months prior to cataract surgery
* CME due to other etiologies such as vein occlusion and diabetes.
* Retinal diseases that preclude evaluation of the macula for edema (e.g., macular hole).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects improving >/= 15 letters (3 lines) of best-corrected distance visual acuity at 18 weeks after initiation of pegaptanib. Distribution of visual acuity changes at 18 weeks after initiation of pegaptanib | 18 weeks after enrollment
Distribution of absolute levels of distance visual acuity at 18 weeks after initiation of pegaptanib | 18 weeks after enrollment
Analysis of time to 15 letter improvement of best-corrected distance visual acuity through 18 weeks after initiation of pegaptanib using a 2-state stochastic model to account for events and recoveries from events | 18 weeks after enrollment

SECONDARY OUTCOMES:
Analysis of decrease in retinal thickness by OCT at 18 weeks after initiation of pegaptanib | 18 weeks after enrollment
Analysis of improvement of fluorescein leakage seen on fluorescein angiography at 18 weeks after initiation of pegaptanib | 18 weeks after enrollment
Additional changes 12 weeks after discontinuation of pegaptanib (6 months after study entry) | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Diana V. Do, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States